CLINICAL TRIAL: NCT06771765
Title: Satiety Promoting Effects of Chia and Hemp Seeds
Brief Title: Soup Meal Satiety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HS69 - Soup Meal Satiety Study
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Obesity Prevention
Keywords: Satiety; Hunger; Fullness; Nutrition
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Lunch Meal (Placebo Comparator): A lunch meal will be provided that is comprised of soup, bread, and a cookie. These items will be made from standard recipes. This arm will be a placebo comparator to meals made with chia seeds or hemp seeds, which may provide extra satiety.
  Interventions: Other: Control (placebo) group
- Chia Enriched Lunch Meal (Experimental): A lunch meal will be provided that is comprised of soup, bread, and a cookie. These items will be made from standard recipes that have been enhanced with chia seeds, which may provide extra satiety compared to the standard recipes in the placebo arm.
  Interventions: Other: Chia Seeds
- Hemp Enriched Lunch Meal (Experimental): A lunch meal will be provided that is comprised of soup, bread, and a cookie. These items will be made from standard recipes that have been enhanced with hemp seeds, which may provide extra satiety compared to the standard recipes in the placebo arm.
  Interventions: Other: Hemp Seeds

INTERVENTIONS:
Other: Chia Seeds — Chia seeds will be added to soup, bread, and a cookie, and these food items will be served as a lunch meal.
  Arms: Chia Enriched Lunch Meal
Other: Hemp Seeds — Hemp seeds will be added to soup, bread, and a cookie, and these food items will be served as a lunch meal.
  Arms: Hemp Enriched Lunch Meal
Other: Control (placebo) group — This intervention is a lunch meal made from standard recipes. This intervention is the placebo control intervention.
  Arms: Control Lunch Meal

SUMMARY:
This study will investigate food ingredients that may provide fullness to healthy adults after a meal. The ingredients will be incorporated into a lunch meal, and measures of hunger and fullness will be evaluated for several hours after the meal. Study subjects must be able to travel to the USDA Nutrition Center in Beltsville Maryland at scheduled times during the study for meals and study measures.

DETAILED DESCRIPTION:
STUDY DESIGN

This study will be a randomized crossover with three treatment periods. Subjects (n=24, approximately equal number of men and women) will be randomly assigned to a treatment sequence.

There will be three 2-day treatment periods separated by a break of ~0-4 weeks, depending on calendar conflicts such as holidays. The treatment period diets will differ in the inclusion of seeds into the recipes on the second day of each period. For all meals on Day 1 and breakfast & lunch on Day 2 of each treatment period, participants will consume a prescribed diet provided by the Beltsville Human Nutrition Research Center. The Day 1 meals and the Day 2 breakfast will be the same for each treatment period (scaled to each participant's intake needs for weight maintenance) so that the participants will be in the same food consumption state the day before the test day. Day 2 lunch will be the treatment meal and will consist of soup, bread, and a dessert item (cookie or brownie). Each of those treatment items (soup, bread, and dessert) will be made one of three ways: (1) by our standard recipe, (2) by our standard recipe modified to include chia seeds, or (3) by our standard recipe modified to include hemp seeds. Dinner on Day 2 will be provided for carry-out and will include a large serving of a dinner entrée, a dessert, and a snack. The Day 2 dinner foods will be provided in excess, and participants will be allowed to eat as much or as little as they like, and they will bring the uneaten portions back to the Beltsville Human Nutrition Research Center the next morning, at which time they will be given a light breakfast, ending the treatment period. The Day 2 dinner items will be weighed before and after the participants eat, and the amount consumed will be recorded and compared across the different recipes to determine if the inclusion of seeds in the recipe promoted satiety. Water will be allowed ad libitum, except that consumption of liquids will not be allowed for the hour before lunch and the hour before dinner on Day 2 of each treatment period.

Participants will complete a series of hunger, fullness, food, and mood related questionnaires during the study.

STUDY PROCEDURES

Controlled feeding intervention: The Beltsville Human Nutrition Research Center will provide all meals to subjects during each 2-day treatment period. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet. For meals on Day 1 and breakfast & lunch on Day 2 of each treatment period, participants will be instructed to eat all foods and only foods provided to them, with the exception of water, coffee, and tea. Coffee and tea intake will be limited to 2 cups per day. Consumption of coffee, tea, and water will be recorded by study subjects. Dinner and snack food for Day 2 of each treatment period will be provided in excess (about 3 times the participants expected calorie needs) and the participants will consume as much or as little of those foods as they like, but they will not be allowed to consume any other foods beyond the foods provided. Alcohol consumption will not be allowed during the intervention.

Body weight: Body weight will be measured at the beginning of each treatment period.

Questionnaires: Participants will be asked to complete a series of questionnaires.

* Participants will complete a questionnaire each study day (6 days total) with questions regarding general health, medications, exercise, and beverage consumption.
* Participants will complete a Three-Factor Eating Inventory on the first morning of the first study session to determine if they are restrained eaters.
* Participants will complete a Positive and Negative Affect Schedule questionnaire before dinner on the second day of each study session to determine if mood states are different among the three study sessions.
* Participants will complete a Visual Analogue Scale assessment of the following subjective feelings at the moment of the assessment: (1) Hunger, (2) Satisfaction, (3) Fullness, (4) Prospective Food Consumption, (5) Desire to Eat something sweet, salty, savory, or fatty. This assessment will be completed on Day 2 of each session, at the following times: immediately before lunch, immediately after lunch, 1 hour after lunch, 2 hours after lunch, 3 hours after lunch, 4 hours after lunch, 5 hours after lunch, and 6 hours after lunch (which will be about 30 minutes after finishing dinner).

Food Intake: Using an analytical scale, Day 2 dinner foods for each participant will be weighed before they are provided to the participants and after the uneaten foods are returned to the Beltsville Human Nutrition Research Center. The weight of the foods will be recorded.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Younger than 25 years
* Known (self-reported) allergy or adverse reaction to study foods
* Women who have given birth during the previous 12 months or who are pregnant/lactating or who plan to become pregnant over the upcoming 6 months (thus during the study period)
* Presence of diabetes, diverticulitis, colitis, celiac disease, Crohn's disease, irritable bowel syndrome, gastrointestinal disease, pancreatic disease
* History of bariatric surgery or other weight control surgery
* Removal of a portion of the stomach or gastrointestinal tract
* Actively trying to gain or lose weight at the time of the study recruitment or planning to gain or lose weight during the study periods
* Diminished sense of taste and/or smell
* Anorexia Nervosa and/or Bulimia
* Smoking, vaping, or use of tobacco products in the past 3 months
* Suspected or known physiological/mechanical GI obstruction
* Use of certain medications or supplements (prescription or over-the-counter) that may interfere with the study objectives
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Feelings of Hunger | 0, 1, 2, 3, 4, 5, and 6 hours post treatment
  Area Under the Curve for Visual Analogue Scale Assessment of Hunger versus Time
Feelings of Satisfaction | 0, 1, 2, 3, 4, 5, and 6 hours post treatment
  Area Under the Curve for Visual Analogue Scale Assessment of Satisfaction versus Time
Feelings of Fullness | 0, 1, 2, 3, 4, 5, and 6 hours post treatment
  Area Under the Curve for Visual Analogue Scale Assessment of Fullness versus Time
Desire to Eat | 0, 1, 2, 3, 4, 5, and 6 hours post treatment
  Area Under the Curve for Visual Analogue Scale Assessment of Desire to Eat versus Time
Dinner Food Intake | 5 hours post intervention
  Weight of food eaten at dinner

CONTACTS AND LOCATIONS:
Overall Officials: Janet Novotny, PhD, Principal Investigator — United States Department of Agriculture (USDA)
Locations (1):
- U.S. Department of Agriculture, Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No